CLINICAL TRIAL: NCT07389395
Title: Comparison of the Effects of Pre-Exercise Instrument-Assisted Soft Tissue Mobilization and Percussion Therapy on Muscle Using a Crossover Design
Brief Title: Grastion and Percussion Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Moxy
Record Dates: First submitted 2025-12-18; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Muscle Fatigue and Muscle Oxygenation
Keywords: Muscle Oxygen Saturation; Muscle Strength; Instrument-Assisted Soft Tissue Mobilization (Graston Technique); Percussion Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instrument-assisted soft tissue mobilization (Active Comparator): With the Graston method, 2 minutes of soft tissue mobilization will be performed on the biceps muscle before the exercise.
  Interventions: Other: Instrument-Assisted Soft Tissue Mobilization (AISM)
- percussion gun (Active Comparator): A percussion gun will be applied to the biceps muscle for 2 minutes before the exercise.
  Interventions: Other: Percussion Therapy
- control (No Intervention): A 2-minute warm-up will be performed without any application.

INTERVENTIONS:
Other: Percussion Therapy — The massage gun will operate at a frequency of 30 beats per second (30 Hz), and percussion therapy will be applied to the muscle for 2 minutes. Percussion therapy will be performed using the device's standard ball head. The force applied by the device will be fixed so that it does not exceed the device's first-stage force setting (approximately 30 pounds). The biceps brachii (dominant arm) will be treated for 2 minutes at 30 Hz, moderate intensity.
  Arms: percussion gun
Other: Instrument-Assisted Soft Tissue Mobilization (AISM) — The arm will be positioned at the edge of the bed in full extension, with the shoulder in 45-degree abduction. The examiner will apply gentle pressure using a 30-degree angled instrument at a rate of 120 strokes/min, aligning the instrument's weight with the fibers of the biceps brachii muscle. The examiner will use a metronome to maintain a consistent pace during treatment, and the instrument angle will be calibrated with a protractor before each subject's treatment. The procedure will last 2 minutes, and baby oil will be used to ensure the instrument moves smoothly over the skin.
  Arms: instrument-assisted soft tissue mobilization

SUMMARY:
The study aims to investigate the effects of percussion therapy and instrument-assisted soft tissue mobilization (AISM), commonly used in clinical settings, on muscle fatigue, maximum muscle strength, pain threshold, and muscle oxygenation.

The study will involve 20 volunteer participants. To achieve the study results, pre-exercise percussion therapy and instrument-assisted soft tissue mobilization (AISM) will be administered using a crossover design.

Results will be measured using a digital dynamometer, a moxy oxygen monitor, and a fatigue questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* Healthy participants
* Sedentary lifestyle as defined by the International Physical Activity Questionnaire (IPAQ) (low physical activity category)
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Upper extremity injury or surgery within the past 6 months
* Presence of skin lesions, wounds, or dermatological diseases at the application site
* Any diagnosed musculoskeletal disorder
* History of cardiovascular, metabolic, or pulmonary disease
* Presence of neurological disorders or cognitive impairment affecting cooperation
* Use of medications affecting neuromuscular function or circulation
* Participation in any upper extremity strength training within the past 3 months
* Contraindications to percussion therapy or instrument-assisted soft tissue mobilization (Graston)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Oxygen Saturation (SmO₂) | "Baseline (30 seconds before exercise)" "During the entire exercise period (from exercise onset to exercise termination)" "Post-exercise (0 to 2 minutes after exercise termination)"
  Oxygen saturation will be measured with the MOXY device. It is an infrared measuring device called "near infrared spectroscopy" that measures oxygen saturation and total hemoglobin in muscle capillaries. The device will be attached to the highest point of the muscle and secured with a black sheath and tape to prevent light exposure.

SECONDARY OUTCOMES:
Muscle Strength | "30, 60, and 90 seconds before the warm-up or intervention" "30, 60, and 90 seconds after the warm-up or intervention" "30, 60, and 90 seconds after exercise"
  Subjects will be seated with the elbow joint flexed to 90°, forearm in supination. They will be asked to contract their muscles in the direction of elbow flexion for 5 seconds, and the physiotherapist will apply force in the opposite direction to prevent movement in the elbow joint. Three measurements will be taken 30 seconds apart, and the average will be recorded.

OTHER OUTCOMES:
Pain Threshold | "120 seconds before the warm-up or intervention" "120 seconds after the warm-up or intervention" "120 seconds after exercise"
  Measurements will be taken at the same point for all participants while the subjects lie supine, with the forearm in full supination at the side of the body and the elbow in full extension. A control trial will be conducted before the measurement, and participants will be instructed to say "OK" as soon as they feel pain
Perceived Fatigue | "Baseline (180 seconds before exercise)" "Post-exercise, immediate (0 minutes)" "Post-exercise (24 hours after exercise termination)" "Post-exercise (48 hours after exercise termination)" "Post-exercise (72 hours after exercise termination)"
  This is a scale used to assess the degree of exertion felt by the participant after exercise. The Borg Scale allows the participant to express the fatigue felt during exercise on a scale of none (6), very light (7-8), light (9-10), fairly light (11-12), somewhat difficult (13-14), difficult (15-16), very difficult (17-18), very very difficult (19), and exhaustion (20)